CLINICAL TRIAL: NCT07231913
Title: Evaluation of the Effectiveness of Emotional Awareness and Communication-Based Intervention Training for Oncology Nurses
Brief Title: Emotional Awareness and Communication Training Effectiveness in Oncology Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, elifcirpanli, MSc Student, Ankara Yıldırım Beyazıt University, Department of Mental Health and Disease Nursing, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07/1398
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Occupational Burnout; Emotional Awareness; Communication Skills
Keywords: Oncology Nurses; Emotional Awareness; Professional Well-being; Psychosocial Training
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups using stratified randomization. The intervention group (n=32) will receive a structured emotional awareness and communication training program over four weeks, consisting of weekly 45-minute face-to-face sessions. The control group (n=32) will receive educational materials in written/digital format after the intervention period. Both groups will be assessed using pre- and post-intervention measures to evaluate emotional awareness, communication skills, and occupational burnout.
Masking Description: This study is open-label. Participants and researchers are aware of group assignments because the intervention involves face-to-face training sessions, which cannot be blinded. Outcome assessments will be conducted using standardized self-report questionnaires. All data will be anonymized during analysis to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive a structured emotional awareness and communication training program over four weeks, with weekly 45-minute face-to-face sessions covering emotional recognition, coping with burnout, effective communication in challenging situations, and personal strategies to prevent burnout.
  Interventions: Behavioral: Structured Emotional Awareness and Communication Training
- Control Group (Other): Participants receive educational materials in written/digital format after the intervention period. No face-to-face training is provided during the study.
  Interventions: Other: Educational Materials

INTERVENTIONS:
Behavioral: Structured Emotional Awareness and Communication Training — Participants in the intervention group will receive a structured training program over four weeks, consisting of weekly 45-minute face-to-face sessions. The program covers:
  Recognizing emotions and emotional awareness Burnout symptoms and healthy coping strategies Challenging conversations and effective communication skills Personal strategies to prevent burnout The training includes interactive presentations, group discussions, and short exercises.
  Arms: Intervention Group
Other: Educational Materials — Participants in the control group will receive written or digital educational materials after the intervention period. No face-to-face training is provided during the study.
  Arms: Control Group

SUMMARY:
This interventional clinical study aims to evaluate whether a structured emotional awareness and communication training program can reduce occupational burnout among oncology nurses. The study will address the following primary questions: Does the intervention lead to a significant increase in nurses' emotional awareness? Does it improve their communication skills in challenging patient and family interactions? Does it reduce their levels of professional burnout? Participants will be recruited from oncology nurses working at Ankara Etlik City Hospital who have been employed in the unit for at least six months and consent to participate. A total of 64 nurses will be randomly assigned to an intervention group (n=32), receiving four weekly face-to-face training sessions over four weeks, or a control group (n=32), receiving educational materials in written/digital format. Data will be collected using pre- and post-intervention assessments with the Maslach Burnout Inventory, the Emotional Requirements Scale, and the Communication Skills Scale for Healthcare Professionals. All data will be anonymized and analyzed to determine the effectiveness of the intervention in enhancing emotional awareness and communication skills and in reducing burnout among oncology nurses.

DETAILED DESCRIPTION:
This interventional study aims to assess the effectiveness of a structured emotional awareness and communication training program in reducing occupational burnout among oncology nurses. The study will be conducted at Ankara Etlik City Hospital Oncology Unit between November 27, 2025, and May 27, 2026. Participants will include 64 nurses who have been working in the unit for at least six months and consent to participate. They will be randomly assigned to an intervention group (n=32) or a control group (n=32) using stratified randomization.

The intervention group will receive four weekly 45-minute face-to-face training sessions covering:

Recognizing Emotions and Emotional Awareness - understanding emotions and their role in professional practice.

Burnout and Healthy Coping Strategies - identifying burnout symptoms and learning adaptive coping mechanisms.

Challenging Conversations and Effective Communication - practicing empathetic listening, reflection, and emotion-focused communication.

Personal Strategies Against Burnout - applying self-care and stress management techniques.

The control group will receive educational materials in written/digital format after the intervention period to ensure ethical compliance. Data will be collected before and after the intervention using the Maslach Burnout Inventory (MBI), the Emotional Requirements Scale, and the Communication Skills Scale for Healthcare Professionals.

All data will be anonymized, and participants' confidentiality will be strictly maintained. Statistical analyses will be performed using International Business Machines (IBM) Statistical Package for the Social Science Statistics (SPSS) 25.0, including independent and paired t-tests and effect size calculations (Cohen's d) to evaluate the intervention's impact on emotional awareness, communication skills, and burnout levels. This study seeks to provide evidence-based strategies to enhance nurses' psychosocial resilience, improve patient care quality, and reduce occupational burnout in high-stress oncology settings.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a nurse in an oncology unit for at least 6 months
* Voluntarily agrees to participate in the study
* Able to attend all training sessions
* Completes both pre-test and post-test questionnaires

Exclusion Criteria:

* Currently on leave or planning to take leave during the study period
* Has received prior structured training related to emotional awareness or communication skills within the past year
* Diagnosed with a severe psychological disorder that may affect participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Burnout Levels of Oncology Nurses | Baseline and 4 weeks after the intervention
  Burnout levels will be assessed using the Maslach Burnout Inventory (MBI) before and 4 weeks after the intervention.

SECONDARY OUTCOMES:
Change in Compassion Fatigue Levels | Baseline and 4 weeks after the intervention
  Compassion fatigue will be evaluated using the Professional Quality of Life Scale (ProQOL) at baseline and 4 weeks after the intervention.
Change in Emotional Awareness and Communication Skills | Baseline and 4 weeks after the intervention
  Emotional awareness and communication skills will be measured using a researcher-developed questionnaire at baseline and 4 weeks after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data collected will be anonymized and used solely for this study. Individual participant data will not be shared outside the research team.